CLINICAL TRIAL: NCT01261455
Title: Prospective Randomized Pilot Study Comparing the Surgical Times Between Inferior Versus Superior Conjunctival Autografts for Primary Pterygia
Brief Title: Prospective Randomized Pilot Study Comparing Inferior Versus Superior Conjunctival Autografts for Primary Pterygia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Allan Slomovic, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB-09-0999A
Record Dates: First submitted 2010-11-22; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-10

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Superior Conjunctival Autograft (Active Comparator): Conjunctival autograft following pterygium excision is taken from superior conjunctival tissue.
  Interventions: Procedure: Location of the autograft taken following pterygium excision
- Inferior Conjunctival Autograft (Experimental): Conjunctival autograft following pterygium excision is taken from inferior conjunctival tissue.
  Interventions: Procedure: Location of the autograft taken following pterygium excision

INTERVENTIONS:
Procedure: Location of the autograft taken following pterygium excision — Following pterygium excision, a conjunctival autograft is taken from either the superior or inferior conjunctiva.

SUMMARY:
The purpose of this study is to determine if there is any difference in the surgical time when the surgery is performed with a graft taken from under the upper lid versus lower lid. The investigators will also be recording the level of pain felt by patients after surgery, any difficulties during or after surgery, and if the pterygium grows back.

ELIGIBILITY:
Inclusion Criteria:

* Primary pterygium (no previous surgeries or radiotherapy) requiring excision due to ocular discomfort or disruption in vision
* Ability to understand the nature of the procedure and to complete all measurement requirements
* Patients must be eligible for either the superior or inferior conjunctival autografts (they must not meet any of the following exclusion criteria)
* Adults (age >18)

Exclusion Criteria:

* Ocular surface disease apart from pterygium (such as severe dry eye, corneal disease, scarring from previous infection, radiotherapy, inflammatory diseases or trauma)
* Patients who have had previous ocular surface surgery
* Patients with glaucoma or those who may need glaucoma surgery in the future
* Contraindications to local anesthetics (such as known allergy)
* Pregnancy (as the risk to the fetus with the use of topical antibiotic drops and local anesthetics are not known)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Time taken to complete the surgical procedure (minutes) | 1 year

SECONDARY OUTCOMES:
Visual Analog Pain Score | 1 week
Recurrence of pterygium | 1 year
Intraoperative and Postoperative Complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Slomovic, MD, Principal Investigator — Toronto Western Hospital, University of Toronto
Locations (1):
- Toronto Western Hospital, University of Toronto, Toronto, Ontario, Canada